CLINICAL TRIAL: NCT05053971
Title: Phase Ib/II Study of ZEN003694 and Entinostat in Advanced and Refractory Solid Tumors
Brief Title: Testing A New Anti-cancer Drug Combination, Entinostat and ZEN003694, for Advanced and Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-09727; NCI-2021-09727 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000033256; 10499 (Other: Yale University Cancer Center LAO); 10499 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-09-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Locally Advanced Pancreatic Carcinoma; Metastatic Pancreatic Carcinoma; Refractory Malignant Solid Neoplasm; Refractory Pancreatic Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Needle; Biopsy, Large-Core Needle; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (entinostat, ZEN003694) (Experimental): PHASE I RUN-IN PERIOD (DAILY DOSING) (NO LONGER USED PER AMENDMENT DATED JUNE 12, 2025): Patients receive ZEN003694 PO QD during days -14 to 1. Patients also undergo core needle biopsy within 30 days prior to starting therapy.
  PHASE I & II COMBINATION TREATMENT (DAILY DOSING) (NO LONGER USED PER AMENDMENT DATED JUNE 12, 2025): Patients receive entinostat PO QW on days 1, 8, 15, and 22, and ZEN003694 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo core needle biopsy on day 1 of cycle 1, and on day 1 of cycle 14.
  PHASE I and PHASE II (INTERMITTENT DOSING): Patients receive entinostat PO on days 1, 8, 15, and 22 of each cycle and ZEN003694 PO QD on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT throughout the study.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Computed Tomography; Procedure: Core Biopsy; Drug: Entinostat

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Core Biopsy — Undergo core needle biopsy
  Other Names: BIOPSY, CORE; CNB; Core Needle; Core Needle Biopsy; Needle Biopsy
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of entinostat and ZEN003694 in treating patients with solid tumors that have spread to other places in the body (advanced) or does not respond to treatment (refractory). Entinostat is in a class of drugs called histone deacetylase (HDAC) inhibitors. It may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. ZEN003694 is an inhibitor of a family of proteins called the bromodomain and extra-terminal (BET). It may prevent the growth of tumor cells that over produce BET protein. This trial aims to test the safety of combination therapy with entinostat and ZEN003694 in treating patients with advanced or refractory solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of BET bromodomain inhibitor ZEN-3694 (ZEN003694) and entinostat in combination in patients with advanced and refractory solid tumors based on dose limiting toxicities (DLTs) of the combination of ZEN003694 and entinostat. (Phase I) II. To determine the overall response rate (ORR) of ZEN003694 and entinostat in advanced/progressive pancreatic cancer. (Phase II)

SECONDARY OBJECTIVES:

I. To describe the safety profile of ZEN003694 and entinostat in advanced and refractory solid tumors. (Phase I) II. To determine the progression-free survival (PFS), duration of response (DOR), and overall survival (OS) of ZEN003694 and entinostat in this patient population. (Phase I) III. To describe the safety profile of ZEN003694 and entinostat in advanced/progressive pancreatic cancer. (Phase II) IV. To determine the progression-free survival (PFS), duration of response (DOR), and overall survival (OS) of ZEN003694 and entinostat in this patient population. (Phase II) V. To assess the effect of ZEN003694 and entinostat therapy on apoptosis, as measured by an apoptosis multiplex immunoassay. (Phase I Daily Dosing of ZEN003694)

EXPLORATORY OBJECTIVES:

I. To assess the effect of ZEN003694 and entinostat therapy on c-MYC and YAP1 as measured by apoptosis immunofluorescence assay. (Phase I Daily Dosing of ZEN003694) II. To assess the effect of ZEN003694 and entinostat therapy on c-MYC and YAP1 as measured by ribonucleic acid (RNA) and protein expression. (Phase I Daily Dosing of ZEN003694) III. To assess the effect of ZEN003694 and entinostat therapy on tumor burden and gene expression patterns as measured by RNA sequencing (RNASeq) on circulating tumor deoxyribonucleic acid (DNA) (ctDNA) specimens. (Phase I Daily Dosing of ZEN003694)

OUTLINE: This is a phase I, dose-escalation study of ZEN003694 in combination with entinostat followed by a phase II study.

PHASE I RUN-IN PERIOD (DAILY DOSING) (NO LONGER USED PER AMENDMENT DATED JUNE 12, 2025): Patients receive ZEN003694 orally (PO) once daily (QD) during days -14 to 1. Patients also undergo core needle biopsy within 30 days prior to starting therapy.

PHASE I & II COMBINATION TREATMENT (DAILY DOSING) (NO LONGER USED PER AMENDMENT DATED JUNE 12, 2025): Patients receive entinostat PO QW on days 1, 8, 15, and 22, and ZEN003694 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo core needle biopsy on day 1 of cycle 1, and on day 1 of cycle 14.

PHASE I and PHASE II (INTERMITTENT DOSING): Patients receive entinostat PO on days 1, 8, 15, and 22 of each cycle and ZEN003694 PO QD on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a) advanced or refractory solid tumor and must meet standard requirements for treatment
* For patients in Phase 2: Patients must have locally advanced, unresectable OR metastatic pancreatic cancer refractory to standard therapy
* For patients with solid tumors, they must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* For patients with solid tumors, they must have received at least one standard of care regimen for metastatic disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ZEN003694, alone or in combination with entinostat, in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin >= 9.0 g/dL (measured within 14 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1,500/mcL (measured within 14 days prior to administration of study treatment)
* Platelets >= 100,000/mcL (measured within 14 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 14 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN (measured within 14 days prior to administration of study treatment)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (measured within 14 days prior to administration of study treatment)
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) test < 1.5 x ULN (measured within 14 days prior to administration of study treatment)
* Albumin > 2.5 g/dL (measured within 14 days prior to administration of study treatment)
* Patients with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Patients must be able to swallow and retain orally administered medication
* Women of childbearing potential must have a negative pregnancy test within 7 days of starting treatment
* The effects of entinostat and ZEN003694 on the developing human fetus are unknown. For this reason and because histone deacetylase inhibitor (HDACi) and BET inhibitor (BETi) agents are known to be teratogenic, women of child-bearing potential and their male partner must agree to use contraception from the time of the screening pregnancy test, continuing for the duration of study participation, and for 3 months after completing the study treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

Exclusion Criteria:

* Patients who have had any anti-cancer therapy within 30 days (or 5 half-lives, whichever is shorter) prior to the first dose of the investigational products
* Patients who have received radiation therapy within 21 days prior to the first dose of the investigational products
* Patients who have a diagnosis of NK cell lymphoma
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, or stable chronic grade 2 toxicities that do not overlap with presumed toxicities of entinostat or ZEN003694
* Patients who are receiving any other investigational agents
* Patients with known untreated or symptomatic brain or leptomeningeal metastases are excluded. Patients with previously treated CNS metastasis may be included provided that they have stable CNS disease for at least 4 weeks (confirmed by imaging) without symptoms and are off corticosteroids (above physiologic dose) for that indication
* Patients with significant malabsorption or nausea and vomiting that would interfere with oral therapies
* Patients with bleeding diathesis or clinically significant bleeding within the prior 6 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat (e.g. medications that have a benzamide structure (tiapride, remoxipride, clebopride) or ZEN003694
* Patients receiving any medications or substances that are strong inhibitors or strong inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows are ineligible. Strong inhibitors or inducers of CYP3A4 and substrates of CYP1A2 must be discontinued at least 7 days prior to the first dose of ZEN003694. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because entinostat is an HDACi and ZEN003694 is a BETi with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with entinostat or ZEN003694, breastfeeding should be discontinued throughout the treatment period and for at least 28 days following the last dose of study treatment if the mother is treated with entinostat or ZEN003694
* Patients with any of the following cardiac criteria:

  * Patients with a corrected QT interval calculated by the Fridericia formula (QTcF) > 450 msec by electrocardiogram (ECG).
  * Concomitant use of any agent known to cause corrected QT interval (QTc) prolongation.
  * Clinically significant conduction abnormalities or arrhythmias.
  * Presence of a cardiac pacemaker or defibrillator with a paced ventricular rhythm limiting ECG analysis.
  * History or evidence of current >= Class II congestive heart failure as defined by New York Heart Association (NYHA).
  * History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 6 months. Subjects with a history of stent placement requiring ongoing antithrombotic therapy (e.g. clopidogrel, prasugrel) will not be permitted to enroll. Clinically significant cardiomegaly, ventricular hypertrophy, or cardiomyopathy
* Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
* Patients with radiation to > 25% of the bone marrow
* Patients who have had a bone-targeted radionuclide within 6 weeks of the first dose of ZEN003694
* Patients who have previously received ZEN003694 or who have been treated with an HDAC inhibitor or investigational BET inhibitor
* Major surgery other than diagnostic surgery, dental surgery or stenting within 4 weeks prior to the first dose of ZEN003694

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase Ib) | Up to 28 days
  The MTD is defined as the highest dose level at which < 33% of the dose cohort (0 of 3 or 1 of 6) experience a dose-limiting toxicity (DLT) in the first cycle. Up to 3 additional patients (maximum enrollment 6) will be added at the MTD level to more fully characterize the safety of the drug combination. If < 33% (2) patients in this expanded cohort experience a DLT, this will be declared the MTD, and thus the phase 2 dose. If 2 or more patients experience a DLT, this dose level will be adopted as the maximum administered dose (MAD) and drop to the dose level immediately below, for the MTD and the phase 2 dose.
Recommended phase 2 dose (RP2D) (Phase Ib) | Up to 28 days
  The RP2D is generally defined as =<1 out of 6 at highest dose level below the maximally administered dose.
Objective response rate (ORR) (Phase II) | Up to 4 weeks post intervention
  Each patient will be assigned one of the following categories: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data). All of the patients who met the eligibility criteria (with the possible exception of those who received no study medication) should be included in the main analysis of the response rate. Patients in response categories 4-9 should be considered to have a treatment failure (disease progression). Thus, an incorrect treatment schedule or drug administration does not result in exclusion from the analysis of the response rate. Precise definitions for categories 4-9 will be protocol specific.

SECONDARY OUTCOMES:
Response rate (RR) in patients with advanced/progressive pancreatic cancer (Phase II) | Up to 4 weeks post intervention
  The exact two-sided 95% confidence intervals (CIs) for the RR will be reported.
Duration of response | Up to 4 weeks post intervention
  The 95% CIs for the duration of response will be reported.
Overall survival | Up to 4 weeks post intervention
  Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on Greenwood's variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. In addition, the 95% CIs for the duration of response will be reported.
Progression free survival | Up to 4 weeks post intervention
  Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on Greenwood's variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. In addition, the 95% CIs for the duration of response will be reported.

OTHER OUTCOMES:
Non-sequencing biomarker analysis | Up to 4 weeks post intervention
  Statistical and bioinformatic data analysis for laboratory non-omics data and clinical data will utilize the following general strategies, as appropriate. For single time-point lab data, tests of hypotheses concerning within-group comparisons will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest. Between-group comparisons will be assessed using either analysis of variance (ANOVA) with adjusted least squares means or Fisher's exact test, for continuous or categorical variables of interest, respectively. For count or binary multiple time-points or correlated data, tests of between-group comparisons will be completed using the generalized estimating equation (GEE) statistical procedure for longitudinal data analysis with multiple observable vectors for the same subject.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm